CLINICAL TRIAL: NCT00580905
Title: Role of Adenosine in the Release of VEGF and Cytokines
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Not enough volunteer recruited before funding could be secured.
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of medicine and pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 070418; CRC-1619
Record Dates: First submitted 2007-12-17; First posted 2007-12-27 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Inflammation
Keywords: Adenosine; Cytokines; Inflammation; VEGF
MeSH Terms: conditions — Inflammation | interventions — Adenosine; Nitroprusside

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): To compare the effects of adenosine at a dose of 80 mcg/kg/min for 30 minutes, Sodium nitroprusside will be used at a dose that produce similar systemic effects (5 mcg/kg/.min)
  Interventions: Drug: Adenosine; Drug: Sodium Nitroprusside
- 2 (Active Comparator): The local effects of adenosine or sodium nitroprusside will be studied in response to microinjection (intradermally) of both drugs. Two microdialysis catheters (CMA 100) will be inserted intradermally in the volar aspect of the forearm after numbing the area with local cold (ice applied in the study area). After 30 minutes,one catheter will be infused with sodium nitroprusside (2microliters/min of a 28 mM solution) and the other with adenosine (2mcl/min of a 100 microM solution) will then be started and continued for 60 minutes. Skin blood flow will be monitored throughout the study with the used of a skin laser Doppler fluxometer mounted adjacent to the area of the microdialysis probe.
  A 2 mm skin biopsy punch will be performed 60 minutes after the end of the infusion.
  Interventions: Drug: Adenosine

INTERVENTIONS:
Drug: Adenosine — IV infusion of adenosine at a dose of 80 mcg/kg/min for 30 minutes.
  Arms: 1
Drug: Sodium Nitroprusside — To compare the effects of adenosine on increasing cytokines, sodium nitroprusside will be infused at 5 mcg/kg/min (a dose expected to produce similar systemic effects to adenosine)
  Arms: 1
Drug: Adenosine — The local effects of adenosine or sodium nitroprusside will be studied in response to microinjection (intradermally) of both drugs. Two microdialysis catheters (CMA 100) will be inserted intradermally in the volar aspect of the forearm after numbing the area with local cold (ice applied in the study area). After 30 minutes,one catheter will be infused with sodium nitroprusside (2microliters/min of a 28 mM solution) and the other with adenosine (2mcl/min of a 100 microM solution) will then be started and continued for 60 minutes. Skin blood flow will be monitored throughout the study with the used of a skin laser Doppler fluxometer mounted adjacent to the area of the microdialysis probe.
  A 2 mm skin biopsy punch will be performed 60 minutes after the end of the infusion.
  Arms: 2

SUMMARY:
The purpose of this study is to extend previous observations in animal models regarding the effects of adenosine in the release of cytokines to human subjects. We intend to accomplish this in two study protocols. In the first we will infuse intravenously adenosine and measure the plasma levels of inflammatory cytokines. In the second one, we will use a microdialysis technique to infuse intradermally small amounts of adenosine and will measure skin blood flow and will take a biopsy to measure levels of mRNA for cytokines.

DETAILED DESCRIPTION:
In Protocol 1 we will infuse adenosine at a dose of 80 mcg/kg/min for 30 minutes while measuring plasma levels of adenosine at different time points, ranging from 30 minutes to 6 hours. Because activation of A2B receptors also mediates the release of inflammatory cytokines, including IL-6, samples will be taken to measure these and other inflammatory/angiogenic cytokines.

In a second protocol, we will administer adenosine intradermically via a microdialysis probe for 30 minutes while we measure the local effect on skin blood flow using laser Doppler techniques. One hour after the end of the infusion we will obtain a skin biopsy from the perfused area for measurement of mRNA for VEGF, IL-8, IL-6 and other cytokines. In addition, we foresee the possibility of further testing looking for and genetic association between angiogenesis and adenosine.

These are proof-of-concept pilot studies. We will study up to 12 subjects in each protocol but an interim analysis will be performed after 6 subjects are studied. This will help us determine if a trend is observed, to perform power calculations, and determine if more extensive studies are warranted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 yr.
* All potential volunteers will have routine blood test to screen for hepatic, renal, and hematological abnormalities.
* Body mass index < 27 Kg/m2 .
* Female volunteers of childbearing potential will undergo HCG pregnancy test at screening and again on the study day.

Exclusion Criteria:

* Pregnancy females
* Subjects unable to give voluntary informed consent
* Subjects on anticoagulant drugs or anemic
* Subjects with a recent medical illness
* Subjects with a history of coronary heart disease
* Subjects with known kidney or liver disease
* Subjects with history of asthma
* Recent (past three days) use of phosphodiesterase type 5 (PDE5) inhibitors (sildenafil, tadalafil or vardenafil)
* History of intolerance to adenosine or nitroprusside
* History of methemoglobinemia
* Use of theophylline products
* Subjects with hematological abnormalities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Plasma levels of cytokines | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States